CLINICAL TRIAL: NCT07033325
Title: Mass Screening for Chagas Disease Among University Entrants as a Strategy to Improve Access to Diagnosis and Treatment in the Province of Salta, Argentina
Brief Title: University-Based Chagas Testing in Salta Province, Argentina
Status: Enrolling by invitation | Type: Observational
Sponsor: Mundo Sano Foundation (Other)
Collaborators: Universidad Nacional de Salta (Other)
Responsible Party: Principal Investigator, Adriana Echazu, Project Director, Mundo Sano Foundation
Other Study IDs: 5/2024-SCRTI-UNSa
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Chagas Disease; Trypanosoma Cruzi Infection; Chronic Chagas Disease
Keywords: Chagas; Chagas Rapid Diagnostic Test; Trypanosoma cruzi; Salta; Argentina
MeSH Terms: conditions — Chagas Disease | interventions — Rapid Diagnostic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum samples will be retained temporarily for the purpose of diagnostic test validation (comparison with recombinant ELISA). No whole blood or DNA will be preserved or extracted. All serum specimens will be properly discarded after testing is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Rapid diagnostic test (RDT) for Trypanosoma cruzi infection. — Rapid diagnostic tests (RDTs) for the detection of Trypanosoma cruzi infection are performed in university facilities, outside of a clinical care setting, using a point-of-care approach. The study population includes adult male and female participants from the university community. This intervention differs from most existing strategies that target exclusively women of reproductive age and/or newborns to control vertical transmission; instead, it focuses on broader population-based screening and linkage to care for chronic infections.
  Other Names: Immunochromatography.; Chagas Rapid Test

SUMMARY:
The goal of this observational study is to improve access to diagnosis and treatment for chronic Trypanosoma cruzi infection among university students of all ages and genders at the National University of Salta (UNSa), Argentina. The main questions it aims to answer are:

* What is the seroprevalence and geographic distribution of T. cruzi infection in UNSa students?
* Can voluntary point-of-care tests performed at university serve as an effective opportunity for timely diagnosis and linkage to care for Chagas disease?

Participants will:

1. Be offered a RDTs (WL Check Chagas, Wiener Lab) during their regular activities in the university.
2. If RDT is positive, be referred to the health system for confirmatory testing and treatment.
3. Receive follow-up support by trained staff via phone. A subgroup of RDT-negative students will have serum samples preserved and analyzed later via ELISA to verify RDT accuracy.

DETAILED DESCRIPTION:
Background and Rationale Chagas disease is a parasitic infection caused by Trypanosoma cruzi, endemic in Latin America and primarily transmitted by triatomine insects. In Argentina, where vector control has reduced transmission, vertical transmission has become the predominant route. The disease often remains asymptomatic for years but can cause serious cardiac and digestive damage during the chronic phase. Specific treatment is available, especially effective if administered early or before pregnancy in women of childbearing age.

Despite the availability of effective therapy, access to diagnosis and treatment remains limited due to both health system and patient-related barriers. The reported prevalence in Salta province is high: around 5% in blood banks and up to 8% among pregnant women.

The Universidad Nacional de Salta (UNSa), with nine campuses across the province, requires all incoming students to complete a medical check-up. This project leverages that existing requirement to offer rapid diagnostic testing (RDT) for T. cruzi, aiming to identify cases early, link positive individuals to care, and indirectly reach affected families.

The study will be implemented by a multidisciplinary team including researchers in medicine, biology, biochemistry, anthropology, and public health, with institutional support from the Universidad Nacional de Salta, Fundación Mundo Sano, and Salta's Ministry of Public Health.

Objectives

Primary Objectives:

1. Increase access to T. cruzi diagnosis and etiological treatment for chronic infections among university students.
2. Prevent congenital transmission of Chagas disease.

Secondary Objectives:

1. Evaluate the use of RDTs in a point-of-care (POC) approach.
2. Determine T. cruzi seroprevalence and geographic distribution among UNSa students.
3. Promote community awareness and knowledge about Chagas disease.
4. Support public health treatment efforts.
5. Assess treatment adherence and safety.
6. Facilitate screening of family members of positive cases.
7. Explore students' knowledge, attitudes, and practices (KAP) regarding Chagas disease.

Methodology

Design:

Implementation research with mixed methods (quantitative and qualitative components).

Study population All incoming students at UNSa in 2024, across all campuses, regardless of age or gender. In addition, other members of the university community (including teachers, administrative staff, and support personnel) who voluntarily choose to participate.

Sites and Estimated Participants:

In 2023, approximately 23,500 students pre-registered, with ~8,000 beginning courses. Campuses are located in Salta Capital, Tartagal, Orán, Metán, Cafayate, Rosario de la Frontera, Santa Victoria Este, San Antonio de los Cobres, and Joaquín V. González. The estimated number of participants is ~5,000.

Procedures

1. Enrollment:

   The Chagas test is offered on a voluntary basis. At the Salta Capital campus, all first-year students are offered the test during their routine medical examination at UNSa, and other members of the university community may also receive the test whenever they visit the university health office. In the regional campuses, testing is carried out through short, intensive Chagas screening campaigns held in university facilities for several weeks during the year, during which any staff or students may participate. Pre-test information is provided, and participants give informed consent.
2. Testing:

   Chagas RDT (WL Check Chagas, Wiener Lab) is performed via fingerstick.
3. Results:

   Participants are informed of results via phone in case of negative results and on-site in case of positive results. Positive cases are referred to the public health system for confirmatory testing (HAI and ELISA) and evaluation (ECG, clinical assessment), and are also contacted by Mundo Sano staff to support follow-up and answer questions.
4. Epidemiological Survey:

   All participants complete a Knowledge, Attitudes, and Practices (KAP) survey, either through an online questionnaire accessed via a QR code or using a printed version when needed.
5. Family and Entomological Surveillance:

   Public health authorities will follow up with family members of positive cases and conduct home vector inspections when applicable.
6. Evaluation of the Diagnostic Test A validation study will be conducted with 100 negative students to compare RDT results with ELISA testing.
7. Treatment Protocol The public health system guarantees confirmation, notification, free drug provision, and medical follow-up. Drugs used: Benznidazole or Nifurtimox.

Treatment adherence, side effects, and outcomes are monitored. Mundo Sano offer telephone or WhatsApp support during treatment.

Data Analysis The analysis will include both quantitative and qualitative components to comprehensively assess the implementation and outcomes of the study.

Quantitative Analysis Data will be collected on the following variables: 1)Demographics: age, sex, current residence, and birthplace. 2) Epidemiological history: including maternal Chagas status, history of blood transfusions, and contact with Chagas vectors. 3)Diagnostic results: including the result of the rapid diagnostic test (RDT) and confirmatory testing (HAI and ELISA). 4) Clinical outcomes: such as treatment status, adherence, adverse effects, and treatment completion among positive cases. 5) Geographic data: for spatial analysis and visualization of case distribution using Geographic Information Systems (GIS).

Descriptive statistics will be used to summarize both continuous and categorical variables. Comparative analyses will be performed using t-tests or Mann-Whitney U tests for continuous variables, and chi-square tests for categorical variables. Associations between key variables will be explored through bivariate and multivariate logistic regression analyses. Geographic distribution of positive cases will be represented using GIS mapping to identify regional patterns of T. cruzi infection within the province.

Data will be managed and analyzed using Microsoft Excel, R statistics, and EPIDAT 4.2.

Qualitative Analysis Qualitative data will be collected through: 1) Pre- and post-treatment Knowledge, Attitudes, and Practices (KAP) surveys. 2) Observations of selected medical consultations (with participant consent). 3) In-depth interviews and extended case studies with a subset of students diagnosed positive. 4) Focus group discussions to explore experiences of participants diagnosed and treated for Chagas. 5) An evaluation of the patient experience with the public health system following diagnosis and referral.

These qualitative methods will provide insight into participants' perceptions of the disease, barriers to care, adherence to treatment, and the overall acceptability of the intervention. Data will be coded and thematically analyzed to identify key patterns and inform future implementation strategies.

Ethical Considerations Approval from Hospital Señor del Milagro and Salta´s Province Bioethics Committee. Informed consent is mandatory. Participation is voluntary and free of charge. Confidentiality is strictly maintained. Results are not a barrier to university entry or employment (per Argentina's National Chagas Law No. 26.281).

ELIGIBILITY:
Inclusion criteria:

* Member of the university community (e.g., student, faculty, administrative staff, or other personnel).
* Aged 18 years or older.
* Of any sex or gender.
* Able and willing to provide informed consent.

Exclusion Criteria:

- Prior confirmed diagnosis of Trypanosoma cruzi infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Salta is a province in northwestern Argentina where Chagas disease remains endemic. While vectorial transmission has declined in recent years due to control efforts, it has not been fully eliminated. Vertical transmission continues to be a major route of infection. Seroprevalence data indicate that 5% of blood donors and 8% of pregnant women in Salta test positive for Trypanosoma cruzi infection.
  The study population includes incoming students at the Nationional University of Salta (UNSa), across its nine campuses located throughout the province. According to UNSa records, in 2023, around 8,000 students began their studies. UNSa is the only public university in Salta, attracting students from across both urban centers and rural areas. First-year students are required to undergo a routine health check, which provides an opportunity for offering Chagas screening. While incoming students are the primary target population, other members of the university are also eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Trypanosoma cruzi infection. | One year.
  Proportion of individuals who tested positive for Trypanosoma cruzi infection among the total number of individuals tested, using Rapid Diagnostic Test (RDT). This outcome reflects the overall frequency of infection within the study population at the time of testing.
Distribution of Trypanosoma cruzi infection. | One year
  Prevalence of T. cruzi infection disaggregated by university campus. This outcome captures the proportion of individuals who tested positive at each participating site, allowing for comparison of infection rates across different geographical locations. The distribution complements the overall prevalence by highlighting site-specific patterns of infection.
Field verification of the RDT | One year
  Diagnostic performance of the RDT for detecting Trypanosoma cruzi infection, assessed in comparison to the reference standard. This outcome reflects the accuracy of the RDT under real-world field conditions in the study population.

SECONDARY OUTCOMES:
Acceptability of the RDT-based testing strategy in a non-health setting | One year
  Level of acceptance of the strategy among participants, staff, and stakeholders involved in the implementation of Trypanosoma cruzi rapid diagnostic testing outside the traditional healthcare setting. This outcome reflects perceptions of appropriateness, comfort, and willingness to engage with the intervention, as reported through surveys, interviews, or informal feedback.
Feasibility of implementing RDT-based testing in a non-health setting | One year
  Extent to which the strategy of offering T. cruzi rapid diagnostic testing in a university or other non-clinical environment can be successfully carried out. This includes assessment of practical aspects such as recruitment, training, workflow integration, space availability, and resource use. The outcome is informed by field observations, implementers' feedback, and process indicators.
Treatment outcomes among participants with confirmed Trypanosoma cruzi infection | 18 months
  This outcome assesses the care cascade following a positive diagnosis, including the number of individuals with confirmed T. cruzi infection who accessed clinical evaluation and received a treatment indication within the public health system. It also includes indicators of treatment initiation, adherence, tolerance (e.g., reported side effects), and completion of therapy. Data are collected through follow-up interviews, clinical records, and coordination with local health services.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Echazu, PhD, Study Director — Mundo Sano Foundation; Ruben O Cimino, PhD, Study Chair — Instituto de Investigaciones de Enfermedades Tropicales, Univeridad Nacional de Salta
Locations (2):
- Argentina (2):
  - Universidad Nacional de Salta, Orán, Salta Province
  - Universidad Nacional de Salta, Salta

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual-level data will be shared, including participants' age, sex, study site (university campus), and results of the rapid diagnostic test (RDT) for Trypanosoma cruzi infection. All data will be de-identified to ensure participant confidentiality, with no personally identifiable information included.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The individual participant data (IPD) will be made available following the completion of the study and the publication of the main results. The anticipated availability period is from December 2025 to June 2026.
Access Criteria: Other researchers will be able to access the IPD information if they need it for scientific purposes and make a formal request describing their objectives.
URL: https://figshare.com/

REFERENCES:
- [Background] Lopez-Albizu C, Danesi E, Piorno P, Fernandez M, Garcia Campos F, Scollo K, Crudo F. Rapid Diagnostic Tests for Trypanosoma cruzi Infection: Field Evaluation of Two Registered Kits in a Region of Endemicity and a Region of Nonendemicity in Argentina. J Clin Microbiol. 2020 Nov 18;58(12):e01140-20. doi: 10.1128/JCM.01140-20. Print 2020 Nov 18. PMID 32938737
- [Background] OPS. Organización Panamericana de la Salud. Guía para el diagnóstico y el tratamiento de la enfermedad de Chagas. Washington, D.C. OPS; 2018. 2018. 1-172 p.
- [Background] Ministerio de Salud de la Nación. Enfermedad de Chagas. Guía para la atención al paciente infectado con Trypanosoma cruzi. 2018. 96 p.
- [Background] WHO Expert Committee. Control of Chagas disease. World Health Organ Tech Rep Ser. 2002;905:i-vi, 1-109, back cover. PMID 12092045